CLINICAL TRIAL: NCT02355067
Title: Social Media Intervention to Teach Parenting for Women With Postpartum Depression
Brief Title: Social Media Intervention for Postpartum Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: The Oscar G. & Elsa S. Mayer Family Foundation (Unknown); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-011491
Record Dates: First submitted 2015-01-30; First posted 2015-02-04 (Estimated); Results first posted 2019-10-02 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-02

CONDITIONS: Postpartum Depression; Parenting
Keywords: parenting; postpartum depression; mothers; infants; depression
MeSH Terms: conditions — Depression, Postpartum; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Media Format (Experimental): Social Media Intervention for women with postpartum depression (PPD) symptoms
  Interventions: Behavioral: Social Media Intervention
- In-Person Format (Active Comparator): Traditional In-Person Intervention for Women with postpartum depression (PPD)
  Interventions: Behavioral: Traditional In-Person Intervention

INTERVENTIONS:
Behavioral: Social Media Intervention — These women will participate in the intervention through the online Facebook group.
  Arms: Social Media Format
Behavioral: Traditional In-Person Intervention — These women will participate in the intervention through a traditional weekly meeting of a group in-person.
  Arms: In-Person Format

SUMMARY:
This study is intended to compare the acceptability and feasibility and explore outcomes related to two different formats of a parenting program for mothers with postpartum depressive symptoms. One version will be a traditional, in-person group format, while the other will be a social media group format. The investigators will also explore the differences in outcomes of both formats, looking at depressive symptoms, parenting sense of competency, and parenting interactions with children.

DETAILED DESCRIPTION:
Postpartum depressive symptoms are common among women following the birth of a child and can adversely impact a mother's ability to care for her child. Evidence-based parent coaching programs have been developed to guide mothers with caring for their infants but do not address the effects of depression on parenting, can be expensive to administer, and are not available in a format that facilitates participation by women with depressive symptoms. We have adapted a previously validated parent coaching intervention, the Parents Interacting with Infants (PIWI) program, for use with depressed parents by inclusion of educational material based on Beardslee's cognitive psycho-educational family model. The program spans 8 weeks, each week focusing on a specific topic. The topics covered are: psychoeducation regarding depression and behavioral activation for coping with high levels of stress, sleep, play, laughter, feeding, temperament, safety, and reading with infants.

We will conduct a pilot randomized controlled trial comparing two versions of the parent coaching program: social media and traditional in-person group formats. We've modified the PIWI program to address barriers to participation through social media format using secret Facebook user groups. We will assess the feasibility and acceptability of the social media program compared to a traditional group format by examining the proportion of subjects who attend group sessions or "like" Facebook sessions. Women who consent to participate in the study will be assigned by randomization to one format or the other in blocks of 20.

Women will complete measures of feasibility and acceptability and measures of depressive symptoms, Beck Depression Inventory-II (BDI-II - Appendix 2) Scale and parenting competence, Parenting Sense of Competency (PSOC - Appendix 3 scales) prior to (time 0) and after the intervention (time 8-12 weeks post enrollment). In addition, mothers and infants in phase III will be videotaped during a 16-minute free play using a standardized measure of parenting interaction (PICCOLO) following completion of the intervention. The measures will provide important information on the effects of parent coaching formats on a new mother's depressive symptoms, her sense of parenting confidence, and her parenting interactions with her infant.

ELIGIBILITY:
Inclusion Criteria:

1. Females
2. 15 years of age or older at the start of the study
3. English speaking
4. Access to the internet via a computer or a smartphone
5. Mother of a child 1-3 months old
6. Edinburgh Postnatal Depression Scale (EPDS) score of 9 or higher
7. Informed consent and HIPAA authorization.

Exclusion Criteria:

1) Have significant suicidal symptoms. Significant suicide risk is defined as current suicidal intent and a plan for suicidal behavior.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2017-11-03 (Actual); Study Completion 2017-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James P Guevara, MD, MPH, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Social Media Format | In-Person Format
Started | 20 | 20
Completed | 12 | 12
Not Completed | 8 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Social Media Format | In-Person Format | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.4 (1.9) | 26.3 (1.8) | 26.3 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 11 | 20
  White | 0 | 1 | 1
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 12 | 24
Beck Depression Inventory II [Mean (Full Range); unit: units on a scale] — The BDI-II is a 21-item self-report tool that measures the severity of depression and includes two subscales: cognitive and somatic. It has been well validated, with scores 14-19 indicating mild depression, 20-28 moderate depression, and 29-63 severe depression. The full range of the BDI-II is 0-64.
  units on a scale | 30.7 [17 to 46] | 25.7 [18 to 35] | 28.2 [17 to 46]
Parenting Sense of Competency [Mean (Full Range); unit: units on a scale] — Measures parental competence on 2 dimensions: Satisfaction and Efficacy. 17-item Likert-scale questionnaire (on a 6 point scale ranging from strongly agree [1] to strongly disagree [6]). Higher scores represent better parenting sense of competency. The full range of the score is 17-102.
  units on a scale | 67.8 [54 to 83] | 78.3 [63 to 97] | 73.0 [54 to 97]

OUTCOME MEASURES:

1. Primary Outcome: Attendance
Description: Percentage of participants who attend each group session or check in online weekly. This is averaged over the course of the 8-week program.
Time Frame: 8 weeks
Measure: Mean (Full Range); unit: percentage of participants
Arm/Group | Social Media Format | In-Person Format
Number analyzed (Participants) | 12 | 12
percentage of participants | 83.3 [67 to 100] | 3.3 [0 to 33]

2. Primary Outcome: Acceptability
Description: Participants report concerning their overall program effects-Satisfaction Questionnaire. The scale ranges from 1-5 with higher values representing higher satisfaction.
Time Frame: 12 weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Social Media Format | In-Person Format
Number analyzed (Participants) | 9 | 4
units on a scale | 4.5 [1 to 5] | 4.5 [1 to 5]

3. Secondary Outcome: Beck Depression Inventory (BDI-II)
Description: The BDI-II is a 21-item self-report tool that measures the severity of depression and includes two subscales: cognitive and somatic. It has been well validated, with scores 14-19 indicating mild depression, 20-28 moderate depression, and 29-63 severe depression. The full range of the BDI-II is 0-64.
Time Frame: 12 weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Social Media Format | In-Person Format
Number analyzed (Participants) | 12 | 8
units on a scale | 20.2 [17 to 40] | 23.3 [14 to 33]

4. Secondary Outcome: Parenting Sense of Competency (PSOC) Scale
Description: The Parenting Sense of Competence scale measures parental competence on two dimensions: Satisfaction and Efficacy. It is a 17 item Likert-scale questionnaire (on a 6 point scale ranging from strongly agree [1] to strongly disagree [6]), with nine questions under Satisfaction and seven under Efficacy. Satisfaction section examines the parents' anxiety, motivation and frustration, while the Efficacy section looks at the parents' competence, capability levels, and problem-solving abilities in their parental role. Higher scores represent better parenting sense of competency. The full range of the score is 17-102.
Time Frame: 12 weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Social Media Format | In-Person Format
Number analyzed (Participants) | 12 | 8
units on a scale | 76.3 [54 to 97] | 73.6 [60 to 92]

ADVERSE EVENTS:
Time Frame: 3 months from enrollment to second study visit
Arm/Group | Social Media Format | In-Person Format
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2015-09-08): https://cdn.clinicaltrials.gov/large-docs/67/NCT02355067/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2015-09-11): https://cdn.clinicaltrials.gov/large-docs/67/NCT02355067/Prot_SAP_001.pdf